CLINICAL TRIAL: NCT05225220
Title: Multimodal Investigation of Post COVID-19 in Females: A Pilot Study
Brief Title: Multimodal Investigation of Post COVID-19 in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Casa Colina Hospital and Centers for Healthcare (Other)
Responsible Party: Principal Investigator, Amy Zheng, Research Scientist, Casa Colina Hospital and Centers for Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#00002372
Record Dates: First submitted 2022-02-02; First posted 2022-02-04 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Post COVID-19; Cognitive Dysfunction
Keywords: Long COVID; Post COVID-19 Syndrome; COVID long-haulers; Brain fog; Anosmia/Hyposmia; Neurological symptoms; EEG; MRI; Genetics; Inflammation; Transcutaneous vagus nerve stimulation; Fatigue; Anxiety; Depression; Cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Post-Acute COVID-19 Syndrome; Mental Fatigue; Anosmia; Neurologic Manifestations; Inflammation; Fatigue; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Transcutaneous Vagus Nerve Stimulation (t-VNS) (Experimental): Participants will receive 60 minutes of t-VNS stimulation every day for 10 consecutive days while wearing a fitness tracker.
  Interventions: Device: Parasym Device (of Parasym Ltd, UK) using Transcutaneous Vagus Nerve Stimulation (t-VNS)

INTERVENTIONS:
Device: Parasym Device (of Parasym Ltd, UK) using Transcutaneous Vagus Nerve Stimulation (t-VNS) — Electrode clip will be placed on the left ear.

SUMMARY:
The purpose of this study is to investigate the effects of transcutaneous vagus nerve stimulation (t-VNS) on Long Covid symptoms in females and to identify factors influencing susceptibility and recovery-particularly in the cognitive domain, as over 80% of long-haulers experience "brain fog".

DETAILED DESCRIPTION:
Long COVID is a post-viral illness estimated to affect 10-30% of COVID-19 patients. Post-COVID symptoms can last for months and affect multiple organs. Major risk factors of long COVID include the female sex and pre-existing anxiety/depression. Because women already have higher rates of anxiety/depression, the combined risks could exacerbate their susceptibility.

Based on the rationale that long COVID symptoms significantly overlap with functions of the vagus nerve, which serves as a conduit between the brain and body, the investigators propose to use non-invasive transcutaneous vagus nerve stimulation (t-VNS) as a novel treatment for long COVID in 20 female participants.

This pilot study will utilize a holistic approach by integrating neuromodulation, neuroimaging, genetics, blood biomarkers, behavioral assessments, and wearable technology to examine the effects of VNS therapy on post COVID-19 symptoms and to identify factors that influence susceptibility and recovery, particularly in the cognitive domain, as over 80% of long-haulers report experiencing "brain fog" (i.e., cognitive disruptions).

ELIGIBILITY:
Inclusion Criteria:

* Biologically female at birth and at time of enrollment
* At least 18 years of age or older
* Experiencing persistent symptoms of brain fog/cognitive impairment beyond 3 months of COVID-19 infection that are not explained by an alternative diagnosis

Exclusion Criteria:

* Not t-VNS compatible (e.g. pacemaker implants)
* Not MRI compatible (e.g. metal implants, claustrophobia)
* Currently pregnant
* Long COVID without cognitive impairment
* History of neurological conditions prior to COVID-19 infection

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be of female sex at birth and at time of study enrollment.
Enrollment: 25 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Change in Flanker Inhibitory Control and Attention Test (Flanker) scores | At baseline, at week 3, and at week 7
  Flanker is a non-verbal NIH Toolbox Cognition Battery assessment that measures both a participant's attention and inhibitory control.
Change in Picture Sequence Memory Test (PSMT) scores | At baseline, at week 3, and at week 7
  PSMT is a non-verbal NIH Toolbox Cognition Battery assessment that measures a participant's episodic memory.
Change in Dimensional Change Card Sort Test (DCCS) scores | At baseline, at week 3, and at week 7
  DCCS is a non-verbal NIH Toolbox Cognition Battery assessment that measures a participant's executive functioning.
Change in Pattern Comparison Processing Speed scores | At baseline, at week 3, and at week 7
  Pattern Comparison Processing Speed is a non-verbal NIH Toolbox Cognition Battery assessment that measures a participant's processing speed.
Change in List Sorting Working Memory scores | At baseline, at week 3, and at week 7
  List Sorting Working Memory is an oral NIH Toolbox Cognition Battery assessment that measures a participant's working memory.

SECONDARY OUTCOMES:
Change in Magnetic Resonance Imaging (MRI) | At baseline and at week 3
  MRI scans will be acquired on a Siemens Magnetom Verio 3T Scanner at Casa Colina Imaging Center to assess structural changes.
Change in resting state Electroencephalograph (EEG) signals | At baseline and at week 3
  Using a 64-channel EEG system, we will perform resting-state EEG recordings to assess power spectral density changes.
Change in blood marker levels | At baseline and at week 3
  Blood markers related to COVID-19, inflammation, brain injury, and neuroplasticity will be analyzed using the Ella automated immunoassay system.
Change in BURNS Anxiety Inventory scores | At baseline, at week 3, and at week 7
  The BURNS Anxiety Inventory is a self-reported rating scale that measures anxiety symptoms.
Change in Becks Depression Inventory (BDI) scores | At baseline, at week 3, and at week 7
  The BDI is a self-reported rating inventory that measures characteristic attitudes and symptoms of depression.
Change in PROMIS Sleep Disturbance scores | At baseline, at week 3, and at week 7
  The PROMIS Sleep Disturbance (8b) is a self-reported measure for perception of sleep quality, depth of sleep, satisfaction with sleep, and perception of difficulty getting and staying asleep.
Change in Fatigue Severity Scale scores | At baseline, at week 3, and at week 7
  The Fatigue Severity Scale is a self-reported 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders.
Change in Sniffin' Sticks olfactory performance | At baseline, at week 3, and at week 7
  The Sniffin' Sticks test (Burghardt®, Wedel, Germany) assesses odor threshold, odor discrimination, and odor identification.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Zheng, PhD, Principal Investigator — Casa Colina Hospital and Centers for Healthcare
Locations (1):
- Casa Colina Hospital and Centers for Healthcare, Pomona, California, United States